CLINICAL TRIAL: NCT00143455
Title: Open Label, Randomised Multicentre Phase III Study Of Irinotecan Hydrochloride (Campto (Registered)) And Cisplatin Versus Etoposide And Cisplatin In Chemotherapy Naive Patients With Extensive Disease - Small Cell Lung Cancer
Brief Title: Study Of Irinotecan Hydrochloride (Campto(R)) And Cisplatin Versus Etoposide And Cisplatin In Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP4174D-3001
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2010-01-21 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PE regimen; Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental)
  Interventions: Drug: Etoposide + cisplatin
- A (Experimental)
  Interventions: Drug: Irinotecan + cisplatin

INTERVENTIONS:
Drug: Etoposide + cisplatin — etoposide 100 mg/m2 days 1, 2 and 3 cisplatin 80 mg/m2 day 1 3 week cycle
  Arms: B
Drug: Irinotecan + cisplatin — irinotecan 65 mg/m2 day 1 and 8 cisplatin 80mg/m2 day 1 3 week cycle
  Arms: A

SUMMARY:
To compare the effects of irinotecan hydrochloride with cisplatin to the "standard" regimen etoposide plus cisplatin on overall survival, in chemotherapy-naive patients with newly diagnosed Extensive Disease-Small Cell Lung Cancer (ED-SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven Small Cell Lung Cancer (SCLC)
* WHO performance status : 0, 1

Exclusion Criteria:

* No previous radiotherapy is allowed except on bone metastases when newly diagnosed. Radiotherapy is not allowed for vena cava syndrome, a stent is recommended ;
* No prior surgery on the primary tumor except for palliative purpose (stent for vena cava syndrome).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2002-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (65):
- Pfizer Investigational Site, Wels, Austria
- Belgium (3):
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
- Czechia (5):
  - Pfizer Investigational Site, Brno-Bohunice
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ostrava - Poruba
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Ústí nad Labem
- Egypt (2):
  - Pfizer Investigational Site, Alexandria
  - Pfizer Investigational Site, Cairo
- France (17):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Bobigny
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Meaux
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Pierre-Bénite
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Brieuc
  - Pfizer Investigational Site, Saint-Etienne
  - Pfizer Investigational Site, Saint-Pierre
  - Pfizer Investigational Site, Villefranche-sur-Saône
  - Pfizer Investigational Site, Villejuif
- Germany (12):
  - Pfizer Investigational Site, Bad Berka
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bovenden-Lenglern
  - Pfizer Investigational Site, Ebensfeld
  - Pfizer Investigational Site, Gauting
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Hemer
  - Pfizer Investigational Site, Löwenstein
  - Pfizer Investigational Site, München
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Perugia
- Netherlands (5):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Maastricht
  - Pfizer Investigational Site, Nieuwegein
- Poland (4):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Otwock
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Warsaw
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Moscow 115 478
  - Pfizer Investigational Site, Saint Petersburg
- Spain (2):
  - Pfizer Investigational Site, Barcelona, BARCELONA
  - Pfizer Investigational Site, Madrid, Madrid
- Switzerland (6):
  - Pfizer Investigational Site, Aarau
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bellinzona
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Ch-4101 Bruderholz
  - Pfizer Investigational Site, Thun
- Taiwan (3):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XRP4174D-3001&StudyName=Study%20Of%20Irinotecan%20Hydrochloride%20%28Campto%28R%29%29%20And%20Cisplatin%20Versus%20Etoposide%20And%20Cisplatin%20In%20Small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of Cohort 1 was terminated early per protocol amendment (29 September 2003). With limited number of subjects in Cohort 1, the efficacy analysis was exploratory. The amendment reduced Irinotecan dose from 80 to 65 mg/m2. With the study powered for Overall Survival in subjects recruited thereafter (Cohort 2) efficacy analysis is reported.
Groups:
- Irinotecan + Cisplatin (Cohort 1): Each chemotherapy cycle was repeated every 21 days (3 weeks) and consisted of : Irinotecan hydrochloride 80 mg/m2 administered intravenously (IV) over 30 - 90 minutes on Day 1 and Day 8 followed by cisplatin 80 mg/m2 administered intravenously (IV) over 30-60 minutes on Day 1.
- Etoposide + Cisplatin (Cohort 1); Etoposide + Cisplatin (Cohort 2): Each chemotherapy cycle was repeated every 21 days (3 weeks) and consisted of: Etoposide 100 mg/m2 administered intravenously (IV) on Day 1, Day 2 and Day 3 followed by cisplatin 80 mg/m2 administered intravenously (IV) over 30-60 minutes on Day 1.
- Irinotecan + Cisplatin (Cohort 2): Each chemotherapy cycle was repeated every 21 days (3 weeks) and consisted of : Irinotecan hydrochloride 65 mg/m2 administered intravenously (IV) over 30 - 90 minutes on Day 1 and Day 8 followed by cisplatin 80 mg/m2 administered intravenously (IV) over 30-60 minutes on Day 1.
Period: Cohort 1
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Started | 39 | 39 | 0 | 0
Received Treatment | 39 | 38 | 0 | 0
Completed | 25 | 22 | 0 | 0
Not Completed | 14 | 17 | 0 | 0
Not completed — Adverse Event | 8 | 4 | 0 | 0
Not completed — Death | 5 | 2 | 0 | 0
Not completed — Progressive Disease | 0 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 0
Not completed — Randomized But Not Treated | 0 | 1 | 0 | 0
Period: Cohort 2
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Started | 0 | 0 | 203 | 204
Received Treatment | 0 | 0 | 202 | 203
Completed | 0 | 0 | 97 | 111
Not Completed | 0 | 0 | 106 | 93
Not completed — Adverse Event | 0 | 0 | 42 | 30
Not completed — No Longer Required Study Treatment | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 4
Not completed — Death | 0 | 0 | 20 | 12
Not completed — Progressive Disease | 0 | 0 | 20 | 27
Not completed — Withdrawal by Subject | 0 | 0 | 13 | 12
Not completed — Other | 0 | 0 | 7 | 6
Not completed — Randomized But Not Treated | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2) | Total
Number analyzed (Participants) | 39 | 38 | 202 | 203 | 482
Age, Customized [Number; unit: participants] — Protocol amendment (29 September 2003) reduced Irinotecan dose from 80 to 65mg/m2. Subjects recruited prior to amendment were referred to as Cohort 1; those afterwards were referred to as Cohort 2.
  participants
    18 to 44 years | 2 | 1 | 11 | 6 | 20
    45 to 64 years | 27 | 24 | 134 | 130 | 315
    > = 65 years | 10 | 13 | 57 | 67 | 147
Sex: Female, Male [Count of Participants; unit: Participants] — Protocol amendment (29 September 2003) reduced Irinotecan dose from 80 to 65mg/m2. Subjects recruited prior to amendment were referred to as Cohort 1; those afterwards were referred to as Cohort 2.
  Participants
    Female | 7 | 7 | 48 | 48 | 110
    Male | 32 | 31 | 154 | 155 | 372

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) for the Full Analysis Population (FAP)
Description: OS was defined as the time from date of randomization to date of death due to any cause. For a subject not expiring, the OS time was censored on the last date of contact that they were known to be alive. The Kaplan-Meier method was used to analyze variables of duration and event associated with possible censoring and estimate the medians survival by treatment groups. The confidence intervals for the medians were calculated using the Brookmeyer and Crowley's method.
Time Frame: Baseline to date of death (every 3 weeks for up to 6 months on study treatment and every 2 months for a minimum of 13 months post study treatment)
Population: FAP = Full analysis population (all treated patients)analyzed in the arm they were assigned by randomization, assuming they had a confirmed small cell lung cancer. The enrollment of Cohort 1 was terminated early per protocol amendment (29 September 2003). With limited number of subjects in Cohort 1, the efficacy analysis was exploratory.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 202 | 203
months |  |  | 10.2177 [8.9692 to 11.6632] | 9.6591 [8.9363 to 11.0719]
Statistical Analysis 1: Comparison: Irinotecan + Cisplatin (Cohort 2) vs Etoposide + Cisplatin (Cohort 2); A non-inferiority test was combined with a superiority test based on a closed testing procedure. The null hypothesis was to be rejected if the lower bound of the 2-sided 95% confidence interval for the hazard ratio (control/test) estimated from a Cox proportional hazards model, with an indicator for the control arm, was less than 0.80; Test type: Superiority or Other; p = 0.0556, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.236, 95% CI [0.995 to 1.536]

2. Secondary Outcome: Number of Subjects With Overall Confirmed Response
Description: Objective disease response = subjects with confirmed complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST). A CR was defined as the disappearance of all target lesions. A PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline to first documentation of confirmed response (every 9 weeks for up to 6 months on study treatment and every 2 months in follow up until progression)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 202 | 203
participants |  |  | 79 | 94
Statistical Analysis 1: Comparison: Irinotecan + Cisplatin (Cohort 2) vs Etoposide + Cisplatin (Cohort 2); Test type: Superiority or Other; p = 0.143, Chi-squared; Odds Ratio (OR) = 1.343, 95% CI [0.905 to 1.993]

3. Primary Outcome: Overall Survival for the Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PP population = a subset of the Cohort 2 FAP. The subjects had to be eligible (subject had no major protocol deviations from inclusion and noninclusion criteria), evaluable for response, without any major protocol deviations during the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 176 | 186
months | 10.5791 [9.2977 to 12.2875] | 9.4292 [8.5092 to 10.1848]
Statistical Analysis 1: Comparison: Irinotecan + Cisplatin (Cohort 2) vs Etoposide + Cisplatin (Cohort 2); Test type: Non-Inferiority or Equivalence — A non-inferiority test was combined with a superiority test based on a closed testing procedure. The null hypothesis was to be rejected if the lower bound of the 2-sided 95% confidence interval for the hazard ratio (control/test) estimated from a Cox proportional hazards model, with an indicator for the control arm, was less than 0.80; p = 0.0110, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.350, 95% CI [1.071 to 1.701]

4. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression. The Kaplan-Meier method was used to analyze variables of duration and event associated with possible censoring and estimate the medians survival by treatment groups. The confidence intervals for the medians were calculated using the Brookmeyer and Crowley's method.
Time Frame: as for outcome 2
Population: FAP = Full analysis population (all treated patients) of Cohort 2 (after the 29 September 2003 protocol amendment), analyzed in the arm they were assigned by randomization, assuming they had a confirmed small cell lung cancer.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 202 | 203
months |  |  | 5.5195 [4.8953 to 6.1437] | 4.8953 [4.8296 to 5.2895]
Statistical Analysis 1: Comparison: Irinotecan + Cisplatin (Cohort 2) vs Etoposide + Cisplatin (Cohort 2); Test type: Superiority or Other; p = 0.0831, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.354, 95% CI [0.961 to 1.908]

5. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from date of randomization to the date of the first documentation of tumor progression. The Kaplan-Meier method was used to analyze variables of duration and event associated with possible censoring and estimate the medians survival by treatment groups. The confidence intervals for the medians were calculated using the Brookmeyer and Crowley's method.
Time Frame: Baseline to date of progression (every 9 weeks for up to 6 months on study treatment and every 2 months for a minimum of 13 months post study treatment until progression)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 202 | 203
months |  |  | 5.3552 [4.9281 to 6.2423] | 6.2423 [5.6838 to 6.7023]
Statistical Analysis 1: Comparison: Irinotecan + Cisplatin (Cohort 2) vs Etoposide + Cisplatin (Cohort 2); Test type: Superiority or Other; p = 0.7544, Cox Proportional Hazard Model; Hazard Ratio (HR) = 0.965, 95% CI [0.771 to 1.208]

6. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 scales include 5 functional scales (physical, role, cognitive, emotional, and social), a global health status/QL scale and 9 symptom scales: nausea and vomiting, pain, fatigue, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. All scales and single-item measures range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, for the global health status/QL represents a high QL (better patient state), and for a symptom scale/item represents a high level of symptomatology/problems (worse patient state).
Time Frame: Baseline, at every cycle (Day -1, Day 1 of cycle before treatment), at the end of the treatment, and every 2 months during follow-up
Population: Data were not analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Tumor Related Symptoms (Pain, Dyspnea, Cough, Hemoptysis, Weight, and the Use of Opioids and Non-Opioids Analgesics)
Description: Improvement of ≥ 1 tumor related symptom = clinical benefit responder. Pain improvement = decrease of ≥ 1 National Cancer Institute (NCI) grade from baseline of ≥ 1 symptom of NCI pain category, without pain symptom worsening. Cough, dyspnea and hemoptysis improvement = decrease of ≥ 1 NCI grade from baseline. Positive weight change ≥ 5 percent gain from baseline. Positive analgesic consumption = change from baseline from opioid to non-opioid category.
Time Frame: Every 3 weeks for up to 6 months on study treatment
Population: Data were not analyzed.
Measure: Number; unit: participants
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Irinotecan + Cisplatin (Cohort 1) | Etoposide + Cisplatin (Cohort 1) | Irinotecan + Cisplatin (Cohort 2) | Etoposide + Cisplatin (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 9/39 | 4/38 | 45/202 | 29/203
Other Adverse Events (participants affected / at risk) | 39/39 | 38/38 | 202/202 | 203/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan + Cisplatin (Cohort 1) (N=39) | Etoposide + Cisplatin (Cohort 1) (N=38) | Irinotecan + Cisplatin (Cohort 2) (N=202) | Etoposide + Cisplatin (Cohort 2) (N=203)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 6
Hand and foot syndrome secondary to sickle cell anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia NOS (Blood and lymphatic system disorders) | 3 | 1 | 10 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 13 | 12
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 6 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac disorder NOS (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiovascular disorder NOS (Cardiac disorders) | 0 | 0 | 1 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1 | 3 | 2
Tachycardia NOS (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular arrhythmia NOS (Cardiac disorders) | 0 | 0 | 0 | 1
Conductive deafness (Ear and labyrinth disorders) | 1 | 1 | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Dry eye NOS (Eye disorders) | 0 | 0 | 1 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual disturbance NOS (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 2 | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis NOS (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 7 | 6
Diarrhoea NOS (Gastrointestinal disorders) | 5 | 1 | 33 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Intestinal obstruction NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 23 | 12
Proctitis NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Vomiting NOS (Gastrointestinal disorders) | 5 | 2 | 22 | 7
Chest pain (General disorders) | 2 | 1 | 11 | 6
Fatigue (General disorders) | 7 | 4 | 25 | 14
General physical health deterioration (General disorders) | 0 | 0 | 14 | 9
Injection site reaction NOS (General disorders) | 0 | 1 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0
Oedema NOS (General disorders) | 1 | 1 | 7 | 4
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Pain NOS (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 10 | 5
Sudden death (General disorders) | 0 | 0 | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Encephalitis herpes (Infections and infestations) | 0 | 0 | 0 | 1
Infection NOS (Infections and infestations) | 2 | 1 | 9 | 6
Lung infection NOS (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia NOS (Infections and infestations) | 0 | 0 | 3 | 1
Respiratory tract infection NOS (Infections and infestations) | 0 | 0 | 1 | 0
Skin fungal infection NOS (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Blood alkaline phosphatase NOS increased (Investigations) | 1 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 5 | 3
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 1 | 9 | 5
Weight decreased (Investigations) | 6 | 0 | 20 | 10
Alkalosis NOS (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 12 | 10
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 5 | 0
General nutrition disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 7 | 8
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1
Dysphonia (Nervous system disorders) | 1 | 1 | 5 | 5
Epilepsy NOS (Nervous system disorders) | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 7 | 5
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Nystagmus NOS (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 3 | 3
Paralysis NOS (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 3 | 0
Syncope (Nervous system disorders) | 0 | 1 | 4 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 8 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 4
Insomnia (Psychiatric disorders) | 2 | 0 | 7 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1 | 0
Incontinence NOS (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure NOS (Renal and urinary disorders) | 0 | 0 | 4 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 25 | 15
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 30 | 22
Expectoration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 4
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 3
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 9 | 6
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Exanthem (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash NOS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 6
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1 | 0
Haematoma NOS (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension NOS (Vascular disorders) | 0 | 0 | 0 | 2
Hypotension NOS (Vascular disorders) | 2 | 0 | 2 | 2
Petechiae (Vascular disorders) | 0 | 0 | 2 | 0
Phlebitis NOS (Vascular disorders) | 0 | 0 | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Convulsions NOS (Nervous system disorders) | 1 | 1 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemorrhage NOS (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan + Cisplatin (Cohort 1) (N=39) | Etoposide + Cisplatin (Cohort 1) (N=38) | Irinotecan + Cisplatin (Cohort 2) (N=202) | Etoposide + Cisplatin (Cohort 2) (N=203)
Leukopenia NOS (Blood and lymphatic system disorders) | 3 | 1 | 21 | 34
Neutropenia (Blood and lymphatic system disorders) | 18 | 18 | 107 | 131
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4 | 26 | 34
Conductive deafness (Ear and labyrinth disorders) | 1 | 5 | 16 | 19
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 17 | 13
Abdominal pain NOS (Gastrointestinal disorders) | 4 | 5 | 27 | 21
Constipation (Gastrointestinal disorders) | 3 | 8 | 41 | 52
Diarrhoea NOS (Gastrointestinal disorders) | 17 | 4 | 113 | 28
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 17 | 17
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 9 | 11
Nausea (Gastrointestinal disorders) | 23 | 22 | 135 | 123
Stomatitis (Gastrointestinal disorders) | 0 | 7 | 21 | 23
Vomiting NOS (Gastrointestinal disorders) | 18 | 18 | 112 | 84
Chest pain (General disorders) | 12 | 12 | 66 | 51
Fatigue (General disorders) | 28 | 27 | 131 | 123
General physical health deterioration (General disorders) | 0 | 0 | 11 | 6
Oedema NOS (General disorders) | 2 | 4 | 29 | 25
Pyrexia (General disorders) | 6 | 0 | 24 | 21
Infection NOS (Infections and infestations) | 1 | 6 | 25 | 32
Blood creatinine increased (Investigations) | 4 | 4 | 32 | 30
Haemoglobin decreased (Investigations) | 7 | 4 | 48 | 50
Weight decreased (Investigations) | 20 | 12 | 83 | 61
Anorexia (Metabolism and nutrition disorders) | 16 | 11 | 81 | 66
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 13 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 13 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 8 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 11 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 10 | 46 | 47
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 10 | 17 | 11
Cholinergic syndrome (Nervous system disorders) | 2 | 0 | 10 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 12 | 12
Dysgeusia (Nervous system disorders) | 3 | 0 | 13 | 8
Dysphonia (Nervous system disorders) | 4 | 4 | 28 | 32
Headache (Nervous system disorders) | 3 | 5 | 35 | 34
Paraesthesia (Nervous system disorders) | 8 | 9 | 54 | 50
Peripheral motor neuropathy (Nervous system disorders) | 1 | 4 | 7 | 13
Anxiety (Psychiatric disorders) | 1 | 3 | 10 | 10
Depression (Psychiatric disorders) | 0 | 2 | 12 | 8
Insomnia (Psychiatric disorders) | 7 | 4 | 27 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 23 | 130 | 130
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 21 | 22 | 134 | 139
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 12 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 21 | 29
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 16 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 22 | 78 | 103
Sweating increased (Skin and subcutaneous tissue disorders) | 0 | 0 | 15 | 20
Hypertension NOS (Vascular disorders) | 0 | 0 | 8 | 11
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 2 | 1 | 0 | 0
Ventricular arrhythmia NOS (Cardiac disorders) | 2 | 1 | 0 | 0
Injection site reaction NOS (General disorders) | 1 | 2 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 2 | 2 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Superior vena caval occlusion (Vascular disorders) | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.